CLINICAL TRIAL: NCT04803149
Title: A Prospective, Multi-center, Randomized, Single-Blind Clinical Trial Comparing COOLIEF* Cooled Radiofrequency to Conventional Radiofrequency Ablation of the Medial Branch Nerves in the Management of Chronic Facetogenic Low Back Pain
Brief Title: Cooled RFA vs Conventional RFA to Manage Chronic Facetogenic Low Back Pain
Acronym: Lumbar CvS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Avanos Medical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 105-20-0006
Record Dates: First submitted 2021-03-12; First posted 2021-03-17 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Chronic Low-back Pain
Keywords: Pain Management; Lumbar facet syndrome; Radiofrequency Ablation; Low Back; Medial Branch Nerves
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant
Masking Description: The study is a participant-blinded trial and deliberate action, utilizing a physical barrier, will be taken to ensure the blind remains intact.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cooled Radiofrequency (Experimental): Cooled radiofrequency energy will be delivered to target medial branch nerves in the lower back to reduce pain
  Interventions: Device: Cooled Radiofrequency
- Conventional Radiofrequency (Active Comparator): Conventional radiofrequency energy will be delivered to target medial branch nerves in the lower back to reduce pain
  Interventions: Device: Conventional Radiofrequency

INTERVENTIONS:
Device: Cooled Radiofrequency — Delivery of energy to ablate sensory nerves via cooled radiofrequency probe
  Other Names: Coolief
  Arms: Cooled Radiofrequency
Device: Conventional Radiofrequency — Delivery of energy to ablate sensory nerves via standard or conventional radiofrequency probe
  Other Names: Standard Radiofrequency
  Arms: Conventional Radiofrequency

SUMMARY:
This study is being conducted to assess the relative effectiveness of radiofrequency neurotomy in subjects with chronic axial low back pain originating in the lumbar facet joints using the COOLIEF* Cooled Radiofrequency Probe as compared to the same procedure conducted using a Standard Radiofrequency Probe.

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized, single-blind comparison study examining the outcomes of subjects with chronic axial low back pain that originates in the lumbar facet joints undergoing a procedure to create a radiofrequency lesion in the medial branch nerves with either Cooled Radiofrequency Ablation (CRFA) or Conventional (Standard) Radiofrequency Ablation (SRFA). Approximately 188 participants from approximately 15 sites will be enrolled into this study, with subjects undergoing either CRFA or SRFA in a 1:1 randomization scheme. Follow-up will be conducted for 12 months post-treatment, with the primary endpoint being completed at month 6. Pain, overall outcome, quality of life, pain medication use, and adverse events will be compared between the two treatment groups to determine success.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 21 years
2. Able to understand the informed consent form and provide written informed consent and able to complete outcome measures.
3. Subjects who have chronic axial (non-radicular) low back pain (at least 3 months) attributed to bilateral L4/L5, L5/S1 lumbar facet joint arthropathy based on clinical evaluation (paraspinal tenderness in the absence of signs and symptoms suggestive of focal neurological deficits) despite conservative treatments, including activity modification, home exercise, protective weight bearing, and/or analgesics (for example, acetaminophen or non-steroidal anti-inflammatory drugs [NSAIDs]).
4. Positive response to dual diagnostic medial branch blocks (defined as a decrease in numeric pain scores of at least 80% for a min of 3 hours for bupivacaine and minimum of 2 hours for lidocaine) using 0.5mL or less of 0.5% bupivacaine and 2% lidocaine, on respective encounters on separate days, at each of the appropriate medial branches.
5. Usual/Average Pain ≥ 6 on an 11-point NRS scale.
6. Analgesics including membrane stabilizers such as Neurontin (gabapentin) and antidepressants for pain, such as Cymbalta (duloxetine), must be clinically stable (defined as stable dosage for ≥ 6 weeks prior to the screening visit) and shall not change during the study without approval of the investigator.
7. Agree to see one physician (study physician) for back pain during the study period.
8. Subjects of child bearing potential must be willing to utilize double barrier contraceptive method for duration of participation.
9. Willingness to comply with the requirements of this protocol for the full duration of the study.

Exclusion Criteria:

1. Evidence of inflammatory arthritis (example, rheumatoid arthritis) or other systemic condition (example; gout, fibromyalgia, MS, Lupus, etc.) that could cause pain.
2. Focal neurologic signs or symptoms.
3. Spinal pathology that may impede recovery such as spina bifida occulta, grade II or higher spondylolisthesis at an affected joint or adjacent level, or significant lumbar scoliosis (sagittal vertical axis angle >5 degrees or Cobb Angle >10 degrees).
4. Suspected mechanical instability based on flexion/extension and/or films at the proposed treatment levels
5. History of prior lumbar fusion or previous lumbar back surgery at the intended treatment levels.
6. Progressive motor deficit, and/or clinical signs of cauda equina or polyradiculopathy.
7. Radiologic evidence of a symptomatic herniated disc or nerve root impingement.
8. Symptomatic moderate or severe foramina or central canal stenosis demonstrating radicular symptoms or neurogenic claudication.
9. Evidence of neuropathic pain affecting the lower back.
10. Intra-articular steroid injection at target levels within 90 days from randomization.
11. Platelet rich plasma (PRP) or stem cells at target levels within 180 days from randomization.
12. Prior lumbar radiofrequency neurotomy of the L3/L4, L4/L5 medial branches and/or L5/S1dorsal ramus.
13. Body mass index (BMI) > 40 kg/m2
14. Extremely thin patients and those with minimal subcutaneous tissue thickness that would not accommodate a radiofrequency lesion of up to 14 mm in diameter to limit the risk of skin burns.
15. Active joint infection or systemic or localized infection at needle entry sites (subject may be considered for inclusion once infection is resolved).
16. Pending or active compensation claim, litigation, or disability remuneration (e.g. disability, worker's compensation, auto injury in litigation or pending litigation).
17. Pregnant, nursing or intent of becoming pregnant during the study period
18. Chronic pain associated with significant psychosocial dysfunction.
19. Poorly controlled severe psychiatric illness or ongoing psychological barriers to recovery, as determined by the investigator.
20. Allergies to any of the medications to be used during the procedures
21. History of uncontrolled coagulopathy, ongoing coagulation treatment that cannot be safely interrupted for procedure, or unexplained or uncontrollable bleeding that is uncorrectable.
22. Identifiable anatomical variability that would materially alter the procedure as described in the protocol.
23. Within the preceding 2 years, subject has suffered from active narcotic addiction, substance, or alcohol abuse.
24. Current prescribed opioid medications greater than 50 morphine equivalent daily opioid dose.
25. Uncontrolled immunosuppression (e.g. AIDS, cancer, diabetes, etc.).
26. Subject currently implanted with pacemaker, stimulator or defibrillator.
27. Participating in another clinical trial/investigation which included therapeutic treatment within 30 days prior to signing informed consent.
28. Subject unwilling or unable to comply with follow up schedule, protocol requirements or procedures.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects whose back pain is reduced by ≥ 50 percent based on the NRS scale at 6 Months | 6 months
  The NRS is an 11-point scale (0 points to 10 points), where 0 points equals "no pain" and 10 points equals "worst pain". There are no sub-scales.
Proportion of subjects experiencing adverse events through 6-months | 6 months

SECONDARY OUTCOMES:
The mean change in SF-36 Physical Functioning (PF) score from baseline to the 6-month visit | 6 months
  Short Form 36-PF - score range = 0 - 100. "0" corresponds to "greatest disability" and "100" indicates "no disability". The means of these scores and their respective standard deviations are reported for each study group
The mean change in Oswestry Disability Index (ODI) score from baseline to the 6-month visit | 6 months
  ODI - score range = 0 - 100. "0" corresponds to "no disability" and "100" indicates the "maximum disability possible". The means of these scores and their respective standard deviations are reported for each study group
The measured Global Perceived Effect scale at the 6-month visit | 6 months
  The Global Perceived Effect is a 7-point scale: 1 point = "worst ever", 2 points = "much worse", 3 points = "worse", 4 points = "not improved but not worse", 5 points = "improved", 6 points = "much improved", 7 points = "best ever". There are no sub-scales.
The mean change in EQ-5D-5L score from baseline to the 6-month visit | 6 months
  This outcome instrument is composed two components. The first component consists of five sub-scales containing five questions each. The point range for each sub-scale is from 1 to 5, with "1" indicating the best study subject condition and "5" indicating the worst study subject condition. Thus, the minimum and maximum scores per sub-scale are 1 and 5, respectively, and such scores for the entire instrument are 5 (best study subject condition) and 25 (worst study subject condition). The sub-scale topics are: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. The second component, EQ-Visual Analog Scale (VAS), has a score range of 0 - 100. "0" corresponds to the "worst imaginable health state" and "100" indicates the "best imaginable health state". The means of these scores and their respective standard deviations are reported for each study group.
The proportion of subjects requiring additional intervention for their back pain during the 6-month period | 6 months

OTHER OUTCOMES:
The proportion of subjects whose back pain is reduced by ≥ 50 percent based on the NRS scale at 12 Months | 12 months
  The NRS is an 11-point scale (0 points to 10 points), where 0 points equals "no pain" and 10 points equals "worst pain". There are no sub-scales.
Proportion of subjects experiencing adverse events through 12 months | 12 months
The mean change in SF-36 Physical Functioning (PF) score from baseline to the 12-month visit | 12 months
  Short Form 36-PF - score range = 0 - 100. "0" corresponds to "greatest disability" and "100" indicates "no disability". The means of these scores and their respective standard deviations are reported for each study group
The mean change in Oswestry Disability Index (ODI) score from baseline to the 12-month visit | 12 months
  ODI - score range = 0 - 100. "0" corresponds to "no disability" and "100" indicates the "maximum disability possible". The means of these scores and their respective standard deviations are reported for each study group
The measured Global Perceived Effect scale at the 12-month visit | 12 months
  The Global Perceived Effect is a 7-point scale: 1 point = "worst ever", 2 points = "much worse", 3 points = "worse", 4 points = "not improved but not worse", 5 points = "improved", 6 points = "much improved", 7 points = "best ever". There are no sub-scales.
The mean change in EQ-5D-5L score from baseline to the 12-month visit | 12 months
  This outcome instrument is composed two components. The first component consists of five sub-scales containing five questions each. The point range for each sub-scale is from 1 to 5, with "1" indicating the best study subject condition and "5" indicating the worst study subject condition. Thus, the minimum and maximum scores per sub-scale are 1 and 5, respectively, and such scores for the entire instrument are 5 (best study subject condition) and 25 (worst study subject condition). The sub-scale topics are: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. The second component, EQ-Visual Analog Scale (VAS), has a score range of 0 - 100. "0" corresponds to the "worst imaginable health state" and "100" indicates the "best imaginable health state". The means of these scores and their respective standard deviations are reported for each study group.
The proportion of subjects requiring additional intervention for their back pain during the 12-month period | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: David Provenzano, Principal Investigator — Pain Diagnostics and Interventional Care
Locations (10):
- United States (10):
  - International Spine & Pain Performance Center, Washington D.C., District of Columbia
  - Millennium Pain Center, Bloomington, Illinois
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Premier Pain Centers, Shrewsbury, New Jersey
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - University Orthopedics Center, Altoona, Pennsylvania
  - Pain Diagnostics and Interventional Care, Sewickley, Pennsylvania
  - University Orthopedics Center, State College, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - The Spine and Nerve Centers of St. Francis Hosptial, Charleston, West Virginia